CLINICAL TRIAL: NCT03754530
Title: A Multi-center, Open Label Study to Determine the Timelines and Effeciency of Icotinib in Combination With Radiation Therapy For NSCLC Patients With Brain Metastases and EGFR Mutation
Brief Title: Icotinib Combined With Radiation Therapy For NSCLC Patients With Brain Metastases and EGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-007-02
Record Dates: First submitted 2018-10-31; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Non-Small Cell Lung Cancer; Brain Metastases
Keywords: NSCLC brain metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — icotinib; Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Icotinib (Experimental): icotinib is administered orally three times per day. Until emerge the progression of the intracranial disease, then is given radiotherapy(>3 with WBRT or <=3 with SRS) after PD
  Interventions: Drug: Icotinib
- Icotinib plus radiation therapy (Experimental): Standard whole brain radiotherapy (WBRT) is given with 30GY/10 times(>3), or SRS(<=3) plus concurrent icotinib, which was administered orally three times per day. Until the disease progresses.
  Interventions: Drug: Icotinib; Radiation: WBRT or SRS

INTERVENTIONS:
Drug: Icotinib — orally three times per day
  Other Names: WBRT or SRS
Radiation: WBRT or SRS — >3 with WBRT;<=3 with SRS
  Other Names: Icotinib
  Arms: Icotinib plus radiation therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of icotinib in combination with radiotherapy for NSCLC patients with brain metastases. The primary endpoint is PFS of intracranial lesions

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is one of the malignant tumors with the highest incidence of brain metastases. Patients with brain metastasis showed poor prognosis and displayed an untreated median survival of only 3-6 months, and most patients died due to the progression of brain metastases. Some research showed that Icotinib alone can improve the efficiency of NSCLC with brain metastases, but there is still unknow about the result about combination with EGFR-TKI and radiotherapy. This study is designed to evaluate the efficacy of icotinib combined with radiotherapy for NSCLC patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of non-small-cell lung cancer (NSCLC) with brain metastases
* Histological or cytological confirmation of EGRF positive sensitive mutation
* Diagnosis of brain metastases on a Gadolinium-enhanced MRI

Exclusion Criteria:

* Previous usage of EGFR-TKI or antibody to EGFR: gefitinib, erlotinib, herceptin, erbitux
* Previous usage of radiation with brain
* CSF or MRI findings consistent with metastases of spinal cord, meninges or meningeal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival of intracranial lesions | 10 months
  Number of participants with progress of intracranial lesions

SECONDARY OUTCOMES:
Progression-free survival | 8 months
  Number of participants with progress of any places in body
Objective response rate of intracranial lesions | 8 weeks
  Number of participants with an objective response. An objective response (OR) was defined as a patient having a best overall response of either complete response (CR) or partial response (PR) according to RECIST, confirmed at least 28 days following the date of the initial response

CONTACTS AND LOCATIONS:
Overall Officials: Li jiancheng, Study Director — Fujian oncology hospital